CLINICAL TRIAL: NCT05962710
Title: FreeStyle Libre 3 Continuous Glucose Monitoring System Confirmation Study
Brief Title: FreeStyle Libre 3 Continuous Glucose Monitoring System
Status: Terminated | Type: Observational
Why Stopped: Study is not required
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC-US-VAL-22221
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: FreeStyle Libre 3 — FreeStyle Libre 3 Continuous Glucose Monitoring System

SUMMARY:
The purpose of this study is to characterize the FreeStyle Libre 3 Continuous Glucose Monitoring System performance with respect to YSI reference venous plasma sample measurements.

DETAILED DESCRIPTION:
This is a pivotal, non-randomized, single arm, multi-center, prospective, nonsignificant risk study to evaluate the FreeStyle Libre 3 Continuous Glucose Monitoring System accuracy and safety. Up to 80 adult subjects (18 years of age or older) and up to 80 pediatric subjects (2-17 years of age) subjects will be enrolled at up to six (6) clinical research sites in the United States. Each subject will wear two sensors for 15 days.

Interstitial glucose readings from each Sensor will be obtained with a corresponding smart phone. Subjects will do up to six (6) scheduled visits to the clinical study site, including the Enrollment/Screening Visit (Visit 1). Based on the subjects' age and/or weight, subjects will have up to three (3) in- clinic visits during which intravenous blood draws and YSI reference testing will occur.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 2 years of age.
2. Subject must have type 1 or type 2 diabetes.
3. Subject must require insulin therapy through an insulin pump and/or multiple daily insulin injections or inhalations (at least 3 daily).
4. Subject must be able to read and understand English.
5. In the investigator's opinion, the subject must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
6. At the time of enrollment, subject must be available to participate in all study visits.
7. For subjects age 2 to 5: willing to allow medical personnel to perform up to 16 capillary fingersticks to allow for capillary blood samples to be obtained per the study protocol.
8. For subjects age 6 and older: willing to allow medical personnel to insert an IV catheter in the arm to allow for venous blood samples to be obtained per the study protocol.
9. Subjects aged 18 years and older must be willing and able to provide written signed and dated informed consent.
10. Subjects aged 17 years and younger must have a parent, guardian or legally authorized representative willing and able to provide written informed consent.
11. Subjects aged 7 - 17 years must be willing and able to provide written signed and dated informed assent.

    Exclusion Criteria:
12. Subjects age 18 and older: Subject is known to be pregnant, attempting to conceive or is not willing and able to practice birth control during the study duration (applicable to only to female subjects age 18 and older).
13. Subjects age 17 and younger: Subject is known to be pregnant or becomes pregnant during the study (only applicable to female subjects age 17 years and younger)
14. Subject has known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
15. Subject has extensive skin changes/diseases at the proposed application sites that could interfere with device placement or the accuracy of interstitial glucose measurements. Such conditions include, but are not limited to extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, dermatitis herpetiformis, skin lesions, redness, infection or edema.
16. Subject is currently participating in another clinical trial.
17. Subject has donated blood within 60 days prior to the beginning of the study activities.
18. For subjects aged 6 years and older: subject has a hemoglobin (Hb) level that is 10% or more below the normal range (for reference the low end of the normal range for Hb for adult males is 12.6 g/dL and for adult females is 11.7 g/dL1; for pediatric males and pediatric females aged 6 - 9 years it is 11.5 g/dL1; for pediatric males and pediatric females aged 10 - 12 it is 12.0 g/dL1; for ; for pediatric males aged 13 - 14 it is 12.0 g/dL and pediatric females aged 13 - 14 it is 11.5 g/dL1; and for pediatric males and pediatric females aged 15 - 17 it is 11.7 g/dL1)
19. Subject has a known concomitant medical condition which, in the opinion of the investigator, could present a risk to the safety or welfare of the subject or study staff.
20. Subject has X-ray, MRI, CT or diathermy appointment scheduled during the period of study participation, and the appointment cannot be rescheduled for a time before study participation starts or after study participation ends.
21. Subject is unsuitable for participation due to any other cause as determined by the investigator.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric subjects with type 1 or type 2 diabetes requiring either prandial rapid acting insulin (administered via injection or inhalation) or continuous subcutaneous insulin infusion (CSII).
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
System Performance | 46 days
  System Performance will be characterized with respect to YSI reference venous plasma measurements

CONTACTS AND LOCATIONS:
Overall Officials: Shridhara A Karinka, PhD, Study Director — Abbott Diabetes Care
Locations (4):
- United States (4):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Rocky Mountain Diabetes & Osteoporosis Center, Idaho Falls, Idaho
  - Diabetes and Glandular Disease Clinic, San Antonio, Texas
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: Undecided